CLINICAL TRIAL: NCT02749136
Title: Phase 2 Study of Neoadjuvant Modified FOLFIRINOX in Patients With Borderline Resectable Pancreas Adenocarcinoma
Brief Title: Neoadjuvant Modified FOLFIRINOX in Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Baek-Yeol Ryoo, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AsanONCHBP-2015-001
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Borderline resectable; Neoadjuvant chemotherapy; FOLFIRINOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perioperative chemotherapy (Experimental): * Preoperative mFOLFIRINOX, every 2 weeks, 8 cycles
  * Postoperative gemcitabine, every 4 weeks, 3-6 cycles
  Interventions: Drug: Preoperative modified FOLFIRINOX and postoperative gemcitabine

INTERVENTIONS:
Drug: Preoperative modified FOLFIRINOX and postoperative gemcitabine — * Preoperative mFOLFIRINOX, every 2 weeks, 8 cycles
    * Oxaliplatin IV 85 mg/m2 Day (D) 1
    * Irinotecan IV 180 mg/m2 D1
    * 5-FU continuous IV infusion 2,400 mg/m2 over 46 hours D1-2
    * Leucovorin IV 400 mg/m2 D1
  * Postoperative gemcitabine, every 4 weeks, 3-6 cycles - Gemcitabine 1,000 mg/ m2 D1, 8, and 15

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy outcomes of neoadjuvant modified FOLFIRINOX and postoperative gemcitabine in patients with borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related death worldwide. The 5-year survival rate in overall patients is less than 6% due to late clinical manifestation and the systemic nature of the disease at presentation. Even in patients with resectable disease, estimated 5-year survival rates after resection are between 15% and 20%. Traditionally, resection alone is regarded as inadequate for cure. Therefore, systemic and/or combined chemotherapy and radiotherapy have been used as preoperative or postoperative therapy.

Neoadjuvant treatment offers several theoretical advantages over an initial resection. Early delivery of systemic therapy for all patients which might lead to the higher rates of negative margin resection rate, and enhanced patient selection for surgery. Although neoadjuvant treatment has been established as a standard of care for resectable or locally advanced disease of breast, gastric, and rectal cancers, the role of neoadjuvant treatment in patients with pancreatic cancer is not clear at present.

There is no global consensus on the management of patients with borderline resectable pancreatic cancer. If initially resected, postoperative adjuvant chemotherapy or chemoradiotherapy is standard. However, there is no standard regimen for neoadjuvant chemotherapy for pancreatic cancer. Recent pivotal phase 2/3 trial has demonstrated that FOLFIRINOX improved the response rates and survival outcomes of patients with metastatic pancreatic cancer compared to gemcitabine.

Because of higher response rates (about 30%) with FOLFIRINOX, this regimen is now widely investigated in the neoadjuvant setting. Therefore, investigators hypothesize that neoadjuvant FOLFIRINOX may enhance the outcomes of patients with borderline resectable pancreatic cancer. This study will assess the feasibility and efficacy outcomes of neoadjuvant modified FOLFIRINOX and postoperative gemcitabine in patients with borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years and older
* Cytologically or histologically confirmed adenocarcinoma of the pancreas
* Met the NCCN criteria for borderline resectable disease (assessed at Aug 23rd, 2015)
* No previous chemotherapy or radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 1
* Adequate bone marrow function as defined by platelets ≥ 100 x 109/L and neutrophils ≥ 1.5 x 109/L
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal (ULN)
* Adequate hepatic function with serum total bilirubin < 2 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other non life-threatening cancer (i.e., prostate or thyroid cancer) except where treated with curative intent > 5 years previously without evidence of relapse
* Written informed consent to the study

Exclusion Criteria:

* No potentially resectable disease or no metastatic disease
* Locally advanced unresectable disease according to the NCCN criteria
* Histologically confirmed adenosquamous carcinoma
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Last dose of radiotherapy received within 4 weeks before the start of study treatment, excluding palliative radiotherapy
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Female subjects who are pregnant or lactating, or males and females of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy from 2 weeks before receiving study drug until 3 months after receiving the last dose of study drug. A highly effective method of contraception is defined as having a low failure rate (< 1% per year) when used consistently and correctly.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
1-year progression-free survival (PFS) rate | 1 year
  PFS rate at 1 year

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  Median PFS
Overall survival (OS) | 3 years
  Median OS
Macroscopic complete resection rate | 5 months
  The rate of no gross residual disease after surgery
Response rate | 4 months
  Response rate defined by Response Evaluation Criteria in Solid Tumor version 1.1
Toxicity profile | 1 year
  Adverse events graded by National Cancer Institute Common Terminology Criteria version 4.03
Biomarker analysis | 3 years
  Blood-based biomarker analysis for the correlation with response rate, progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Baek-Yeol Ryoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz MH, Marsh R, Herman JM, Shi Q, Collison E, Venook AP, Kindler HL, Alberts SR, Philip P, Lowy AM, Pisters PW, Posner MC, Berlin JD, Ahmad SA. Borderline resectable pancreatic cancer: need for standardization and methods for optimal clinical trial design. Ann Surg Oncol. 2013 Aug;20(8):2787-95. doi: 10.1245/s10434-013-2886-9. Epub 2013 Feb 23. PMID 23435609
- [Background] O'Reilly EM, Perelshteyn A, Jarnagin WR, Schattner M, Gerdes H, Capanu M, Tang LH, LaValle J, Winston C, DeMatteo RP, D'Angelica M, Kurtz RC, Abou-Alfa GK, Klimstra DS, Lowery MA, Brennan MF, Coit DG, Reidy DL, Kingham TP, Allen PJ. A single-arm, nonrandomized phase II trial of neoadjuvant gemcitabine and oxaliplatin in patients with resectable pancreas adenocarcinoma. Ann Surg. 2014 Jul;260(1):142-8. doi: 10.1097/SLA.0000000000000251. PMID 24901360
- [Background] Heinemann V, Haas M, Boeck S. Neoadjuvant treatment of borderline resectable and non-resectable pancreatic cancer. Ann Oncol. 2013 Oct;24(10):2484-2492. doi: 10.1093/annonc/mdt239. Epub 2013 Jul 12. PMID 23852311
- [Background] Lee JL, Kim SC, Kim JH, Lee SS, Kim TW, Park DH, Seo DW, Lee SK, Kim MH, Kim JH, Park JH, Shin SH, Han DJ. Prospective efficacy and safety study of neoadjuvant gemcitabine with capecitabine combination chemotherapy for borderline-resectable or unresectable locally advanced pancreatic adenocarcinoma. Surgery. 2012 Nov;152(5):851-62. doi: 10.1016/j.surg.2012.03.010. Epub 2012 Jun 6. PMID 22682078
- [Background] Heestand GM, Murphy JD, Lowy AM. Approach to patients with pancreatic cancer without detectable metastases. J Clin Oncol. 2015 Jun 1;33(16):1770-8. doi: 10.1200/JCO.2014.59.7930. Epub 2015 Apr 27. PMID 25918279
- [Background] Oettle H, Post S, Neuhaus P, Gellert K, Langrehr J, Ridwelski K, Schramm H, Fahlke J, Zuelke C, Burkart C, Gutberlet K, Kettner E, Schmalenberg H, Weigang-Koehler K, Bechstein WO, Niedergethmann M, Schmidt-Wolf I, Roll L, Doerken B, Riess H. Adjuvant chemotherapy with gemcitabine vs observation in patients undergoing curative-intent resection of pancreatic cancer: a randomized controlled trial. JAMA. 2007 Jan 17;297(3):267-77. doi: 10.1001/jama.297.3.267. PMID 17227978
- [Background] Neoptolemos JP, Stocken DD, Bassi C, Ghaneh P, Cunningham D, Goldstein D, Padbury R, Moore MJ, Gallinger S, Mariette C, Wente MN, Izbicki JR, Friess H, Lerch MM, Dervenis C, Olah A, Butturini G, Doi R, Lind PA, Smith D, Valle JW, Palmer DH, Buckels JA, Thompson J, McKay CJ, Rawcliffe CL, Buchler MW; European Study Group for Pancreatic Cancer. Adjuvant chemotherapy with fluorouracil plus folinic acid vs gemcitabine following pancreatic cancer resection: a randomized controlled trial. JAMA. 2010 Sep 8;304(10):1073-81. doi: 10.1001/jama.2010.1275. PMID 20823433
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Christians KK, Tsai S, Mahmoud A, Ritch P, Thomas JP, Wiebe L, Kelly T, Erickson B, Wang H, Evans DB, George B. Neoadjuvant FOLFIRINOX for borderline resectable pancreas cancer: a new treatment paradigm? Oncologist. 2014 Mar;19(3):266-74. doi: 10.1634/theoncologist.2013-0273. Epub 2014 Feb 25. PMID 24569947
- [Derived] Lim DH, Yoon H, Kim KP, Ryoo BY, Lee SS, Park DH, Song TJ, Hwang DW, Lee JH, Song KB, Kim SC, Hong SM, Hyung J, Yoo C. Analysis of Plasma Circulating Tumor DNA in Borderline Resectable Pancreatic Cancer Treated with Neoadjuvant Modified FOLFIRINOX: Clinical Relevance of DNA Damage Repair Gene Alteration Detection. Cancer Res Treat. 2023 Oct;55(4):1313-1320. doi: 10.4143/crt.2023.452. Epub 2023 May 4. PMID 37139665
- [Derived] Yoo C, Lee SS, Song KB, Jeong JH, Hyung J, Park DH, Song TJ, Seo DW, Lee SK, Kim MH, Lee SS, Kim JH, Jin HS, Park JH, Hwang DW, Lee JH, Lee W, Chang HM, Kim KP, Ryoo BY, Kim SC. Neoadjuvant modified FOLFIRINOX followed by postoperative gemcitabine in borderline resectable pancreatic adenocarcinoma: a Phase 2 study for clinical and biomarker analysis. Br J Cancer. 2020 Aug;123(3):362-368. doi: 10.1038/s41416-020-0867-x. Epub 2020 May 20. PMID 32433600